CLINICAL TRIAL: NCT01129687
Title: Multicenter Prospective Analysis of Treatment Outcome in Patients With Large Acoustic Neuromas
Brief Title: Subtotal Resection of Large Acoustic Neuromas With Possible Stereotactic Radiation Therapy
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: University of Cincinnati (Other); Baylor College of Medicine (Other); Weill Medical College of Cornell University (Other); University of Iowa (Other); University of Texas (Other); George Washington University (Other); Indiana University (Other); Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Ashkan Monfared, Principal Investigator, George Washington University
Other Study IDs: SU-03052010-5142
Record Dates: First submitted 2010-03-10; First posted 2010-05-25 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Neuroma, Acoustic
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Microsurgery; Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ANSRS group: Patients qualifying for the study.
  Interventions: Procedure: Microsurgery; Procedure: Stereotactic radiation therapy

INTERVENTIONS:
Procedure: Microsurgery — Patient would under to total, near-total, or subtotal resection of tumor
Procedure: Stereotactic radiation therapy — Patient who has sign of growth of tumor remnant would undergo this treatment

SUMMARY:
The investigators study is to investigate safety and efficacy of performing a planned incomplete removal of large acoustic neuroma tumors to decrease surgical morbidity and yet avoid tumor recurrence by post-operative radiation therapy.

DETAILED DESCRIPTION:
The current standard treatment of a large tumor of the balance nerve (acoustic neuroma or vestibular schwannoma) is surgical resection. Complete removal of such tumor is associated with significant risks of hearing loss and facial paralysis whereas incomplete removal of the tumor is associated with significant risks of regrowth. Stereotactic radiation is a well accepted therapy aiming at stopping the growth of smaller acoustic neuromas before their sizes become large enough to cause problems. The purpose of our study is to determine whether the combination of subtotal resection followed by stereotactic radiation of the remnant can control large acoustic neuromas without the significant risks associated with complete resection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with acoustic neuromas the widest diameter of 2.5 cm or larger at the cerebellopontine angle are eligible for this trial.
* Patients that are deemed good surgical candidates based on age, general health, genetic predispositions, and hearing in contralateral side would be included as the subjects of this trial.
* Although we would include patients with neurofibromatosis II in this trial, considering their genetic predisposition for recurrence, we would analyze their outcome as a separate group.

Exclusion Criteria:

* Patients who have received any form of treatment of their acoustic neuromas prior to enrollment in the study including surgery or radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with large acoustic neuromas measuring 2.5cm in longest dimension in the cerebellopontine angle.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2005-03; Primary Completion 2022-05-08 (Actual); Study Completion 2022-05-08 (Actual)

PRIMARY OUTCOMES:
Need for stereotactic radiation therapy should tumor remnant grow on annual MRI's | 10 years

SECONDARY OUTCOMES:
Facial nerve function measured on House-Brackmann scale | 10 y

CONTACTS AND LOCATIONS:
Overall Officials: Ashkan Monfared, MD, Study Director — George Washington University; Robert K Jackler, MD, Study Director — Stanford University
Locations (9):
- United States (9):
  - Stanford University School of Medicine, Stanford, California
  - George Washington University, Washington D.C., District of Columbia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Louisiana State University, Baton Rouge, Louisiana
  - Weill Cornell Medical College, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas